CLINICAL TRIAL: NCT03655652
Title: Preoperative Progression of fovea-on Retinal Detachment
Brief Title: Preoperative Progression of Retinal Detachment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Mark Alberti, Principal Investigator, Glostrup University Hospital, Copenhagen
Other Study IDs: H-17015584
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Retinal Detachment
Keywords: positioning
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients are required to position prior to retinal detachment surgery. We seek to see whether there is a correlation between the performed positioning and retinal detachment progression/regression in fovea-on retinal detachment patients.

ELIGIBILITY:
Inclusion Criteria:

* fovea-on retinal detachment
* informed consent

Exclusion Criteria:

* previous retinal detachment surgery
* >14 days of retinal detachment symptoms
* split-fovea retinal detachment
* other retinal disease with influence on retinal biomechanics/elasticity (proliferative diabetic retinopathy, wet AMD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a fovea-on retinal detachment referred to Rigshospitalet - Glostrup Department of Ophthalmology.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Retinal detachment progression/regression | 1-72 hours
  Measured by OCT

SECONDARY OUTCOMES:
Positioning | 1-72 hours
  Measured by device

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Rigshospitalet - Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided